CLINICAL TRIAL: NCT00078221
Title: Rheopheresis Blood Filtration Study for the Treatment of Dry Age-Related Macular Degeneration (AMD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OccuLogix (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AMD-02-99
Record Dates: First submitted 2004-02-20; First posted 2004-03-01 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2005-12

CONDITIONS: Macular Degeneration
Keywords: Dry AMD; Age-related Macular Degeneration; Rheopheresis
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Device: Rheopheresis blood filtration

SUMMARY:
AMD is a progressive disease of the retina which is nourished by a network of tiny blood vessels. There is evidence to suggest that the flow of nutrients to the retina is impaired in patients with AMD. Rheopheresis blood filtration uses blood filters that deplete excesses of large proteins, fats and other substances from the blood, improving blood flow to the macula, potentially improving vision.

ELIGIBILITY:
* Age 50-85
* Diagnosis of Dry AMD
* BCVA between 20/32 and 20/125 in at least one eye
* Numerous large plaques (soft drusen)
* No history of HIV, Hepatitis B or C
* Elevation of certain blood factors, such as total cholesterol, fibrinogen, and IgA

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 1999-08; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Irving Siegel, MD, Study Director — OccuLogix
Locations (8):
- United States (7):
  - Retina Vitreous Associates, Beverly Hills, California
  - Aran Eye Associates, Coral Gables, Florida
  - Retina Health Care, Fort Myers, Florida
  - UIC Eye Center, Chicago, Illinois
  - Macula Care, New York, New York
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Associated Retinal Consultants, Bala-Cynwyd, Pennsylvania
- W. Bradley Kates, MD, Oakville, Ontario, Canada

REFERENCES:
- [Background] Pulido JS; Multicenter Investigation of Rheopheresis for AMD (MIRA-1) Study Group. Multicenter prospective, randomized, double-masked, placebo-controlled study of Rheopheresis to treat nonexudative age-related macular degeneration: interim analysis. Trans Am Ophthalmol Soc. 2002;100:85-106; discussion 106-7. PMID 12545682
- See also: Related Info — http://www.rheo.com